CLINICAL TRIAL: NCT03865524
Title: Effect Of The Use Of Navigation In The Alignment Obtained When Performing A Total Knee Arthroplasty In Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pedro-José Torrijos-Garrido (Other)
Responsible Party: Sponsor-Investigator, Pedro-José Torrijos-Garrido, Principal Investigator, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAOBE
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis, Knee; Obesity; Arthropathy of Knee
Keywords: Osteoarthritis, Knee; Obesity; Knee replacement; Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, Multicenter, prospective trial with a CE-marked medical device
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Total knee arthroplasty implanted with GPS navigation system.
  Interventions: Device: Total knee arthroplasty implanted with GPS navigation system
- Control (Active Comparator): Total knee arthroplasty implanted with standard guides.
  Interventions: Device: Total knee arthroplasty implanted with standard guides.

INTERVENTIONS:
Device: Total knee arthroplasty implanted with GPS navigation system — Obese patients undergoing Total Knee Arthroplasty, GPS achieved alignment
  Arms: Experimental
Device: Total knee arthroplasty implanted with standard guides. — Obese patients undergoing Total Knee Arthroplasty, alignment achieved by using standard guides
  Arms: Control

SUMMARY:
NAOBE is a randomized, open and prospective clinical trial that evaluates the accuracy to achieve an adequate mechanical axis of the lower extremity in obese patients after total knee replacement.

DETAILED DESCRIPTION:
Randomized, open and prospective clinical trial.

Following the surgical indication for a total knee replacement as treatment for symptomatic osteoarthritis and the confirmation of obesity (BMI equal or greater than 30 Kg/m2 ), patients will be randomly assigned (ratio 1:1) to one of the following treatments:

Control group: Total knee arthroplasty implanted with standard guides . Experimental group: Total knee arthroplasty(TKA) implanted with GPS navigation system Patient (or their legal guardian) must provide/sign the informed consent prior to inclusion in the study.

After the surgery, patients will be followed-up at 6 weeks, 3, 6 and 12 months. At those times, data regarding physical and radiological examinations, pain and functionality and health status questionnaires will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old.
* Written informed consent according to ICH / GCP and Spanish legislation, obtained before any study procedure.
* Patient with a BMI equal to or greater than 30 Kg / m2
* Patients with clinical and radiological criteria of knee osteoarthritis.
* Patients with indication for primary TKA according to medical criteria.

Exclusion Criteria:

* Pregnancy or lactation.
* Inability to give informed consent in the absence of a legal representative.
* Subjects that are participating in a study with medicines or other medical devices.
* Those who show inability to follow the instructions or collaborate during the development of the study.
* If in the opinion of the researcher there are findings in the physical examination, abnormalities in the results of the clinical analyzes or other medical, social or psychosocial factors that could have a negative influence
* Having had a previous surgical procedure on or around the knee in the last 12 months (such as proximal tibial osteotomy, femoral osteotomy, open reduction and internal fixation for a fracture, patellectomy or patellar realignment).
* Need a simultaneous bilateral TKA.
* Have a varus angle or valgus ≥ 15 °.
* Total revision knee arthroplasty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Deviation in a mechanical axis of knees | 12 months
  Proportion of knees after surgery with a mechanical axis with a deviation greater than 3º

SECONDARY OUTCOMES:
Radiological axes (femoral) | 12 months
  Position angle of the femoral component: angle formed between the anatomical axis of the femur and the articular surface of the femoral component of the TKA (α).
Radiological axes (tibial) | 12 months
  Position angle of the tibial component: angle formed between the anatomical axis of the tibia and the proximal surface of the tibial component of the TKA (β).
Surgical procedure time | Week 1
  Surgical time
Admission (hospital) duration | Week 1
  Number of days of the hospital admission
Number of Surgical complications (Intraoperative) | Week 1
  Intraoperative complications
Number of Surgical complications (perioperative) | 1 to 6 weeks
  perioperative complications
Number of Surgical complications (post-operative) | 1-12 months
  postoperative complications

OTHER OUTCOMES:
Knee Society Score Questionaire | 6 weeks-12 months
  KSS Questionaire, developed by the Knee Society, assesses the function of the knee replacement and the functional capabilities of patients after their implantation.
  It has to separate sections ("Knee Score" and "Functional Score") that are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
Range of Motion | 6 weeks-12 months
  The maximum extension and flexion
Visual Analogic Scale for pain | 1-12 months
  VAS measure the intensity of the pain that the patient describes. It consists of a horizontal line of 10 centimeters, with 0cm being "no pain" and 10cm being "extreme pain".

CONTACTS AND LOCATIONS:
Overall Officials: Pedro José Torrijos Garrido, MD, PhD, Principal Investigator — Hospital Universitario Puerta de Hierro
Locations (2):
- Spain (2):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Santa Cristina, Madrid

IPD SHARING:
Plan to Share IPD: No